CLINICAL TRIAL: NCT02465866
Title: A Single-Dose, Four-Period, Four-Treatment, Four-Way Crossover Relative Bioavailability Study of CL-108 Under Fed and Fasted Conditions
Brief Title: A Four-Period, Four-Treatment, Four-Way Relative Bioavailability Study of CL-108 Under Fed and Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charleston Laboratories, Inc (Industry)
Responsible Party: Principal Investigator, Joseph Hazelton, Vice-President, Regulatory Affairs, Charleston Laboratories, Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CLCT-004
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Plasma concentration; Time to plasma concentration; Elimination rate constant; Elimination half life; Area under the curve
MeSH Terms: interventions — hydrocodone tartrate, ibuprofen drug combination; Ultracet; Promethazine; Diphenhydramine

ARMS (4):
- Treatment A: CL-108 (Fasted) (Experimental): CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fasted condition
  Interventions: Drug: CL-108
- Treatment B: CL-108 (Fed) (Experimental): CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fed condition
  Interventions: Drug: CL-108
- Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) (Active Comparator): Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fasted condition
  Interventions: Drug: Vicoprofen; Drug: Ultracet; Drug: Phenergan
- Treatment D: Vicoprofen, Ultracet and Phenergan (Fed) (Active Comparator): Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fed condition
  Interventions: Drug: Vicoprofen; Drug: Ultracet; Drug: Phenergan

INTERVENTIONS:
Drug: CL-108 — Hydrocodone bitartrate/acetaminophen/promethazine 7.5 mg/325 mg/12.5 mg single dose by mouth
  Arms: Treatment A: CL-108 (Fasted); Treatment B: CL-108 (Fed)
Drug: Vicoprofen — Hydrocodone Bitartrate and Ibuprofen 7.5 mg/200 mg single dose tablet by mouth
  Arms: Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted); Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Drug: Ultracet — Tramadol HCl/acetaminophen 37.5 mg/325 mg single dose tablet by mouth
  Arms: Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted); Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Drug: Phenergan — Phenergan (Promethazine HCl, USP) 12.5 mg single dose tablet by mouth
  Other Names: Promethazine HCl
  Arms: Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted); Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)

SUMMARY:
This study will compare the relative bioavailability of hydrocodone, acetaminophen, and promethazine in CL-108 (hydrocodone 7.5mg/ acetaminophen 325 mg/ promethazine 12.5 mg) manufactured by Charleston Laboratories, Inc. to hydrocodone in Vicoprofen (hydrocodone 7.5 mg /ibuprofen 200 mg), promethazine 12.5 mg, and acetaminophen in Ultracet (tramadol HCl 37.5 mg/acetaminophen 325 mg) under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Subject's body mass index (BMI) must be between 18 and 30kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110lb)
* Abide by study restrictions
* Acceptable birth control measures
* Ability to attend all study visits
* Vital signs as per protocol
* Willing to consume high calorie meals within designated time frame

Exclusion Criteria:

* Clinically significant medical history
* Clinically significant abnormal findings
* History or presence of allergic or adverse response to hydrocodone, ibuprofen,acetaminophen, any non-steroidal anti-inflammatory drugs (NSAIDs), promethazine, or related drugs.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication
* Has donated blood or plasma within 30 days prior to the first dose of study medication
* Has participated in another clinical trial (randomized subjects only) within 30 days prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty healthy subjects were enrolled in the study.
Groups:
- Sequence 1: ABDC: Treatment A: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fasted condition
  Treatment B: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fed condition
  Treatment D: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fed condition
  Treatment C: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fasted condition
  Dosing in 4 study periods was separated by a 14-day washout period
- Sequence 2: BCAD: Treatment B: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fed condition
  Treatment C: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fasted condition
  Treatment A: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fasted condition
  Treatment D: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fed condition
  Dosing in 4 study periods was separated by a 14-day washout period
- Sequence 3: CDBA: Treatment C: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fasted condition
  Treatment D: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fed condition
  Treatment B: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fed condition
  Treatment A: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fasted condition
  Dosing in 4 study periods was separated by a 14-day washout period
- Sequence 4: DACB: Treatment D: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fed condition
  Treatment A: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fasted condition
  Treatment C: Vicoprofen 7.5 mg/200 mg + Ultracet 37.5 mg/325 mg + Phenergan 12.5 mg single dose tablets by mouth under fasted condition
  Treatment B: CL-108 single dose tablet (7.5 mg/325 mg/12.5 mg) by mouth under fed condition
  Dosing in 4 study periods was separated by a 14-day washout period
Period: Period 1
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 1: Washout (14 Days)
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 2: Washout (14 Days)
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 5 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Period 3: Washout (14 Days)
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 4 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 4 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 4: Washout (14 Days)
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 4 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Subjects
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.85 (17.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Black or African American | 2
  White | 17
Region of Enrollment [Number; unit: participants]
  United States | 20
Height [Mean (Standard Deviation); unit: cm] | 163.15 (10.49)
Weight [Mean (Standard Deviation); unit: kg] | 67.83 (10.72)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 25.43 (2.80)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration (Cmax) in Plasma Determined Directly From Individual Concentration-time Data
Description: Cmax of CL-108 and Vicoprofen + Ultracet + Phenergan were measured in the plasma (the liquid component of the blood in which the blood cells are suspended) in samples collected up to 48 hours post-dose.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: Intended to treat (ITT) population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
ng/mL
  Hydrocodone | 20.0 (5.48) | 17.9 (5.80) | 18.4 (5.62) | 17.5 (3.63)
  Acetaminophen | 4.71 (1.49) | 3.27 (1.00) | 5.02 (1.66) | 3.03 (0.919)
  Promethazine (Number of Participants=19,19,20,19) | 4.79 (3.75) | 3.66 (2.16) | 4.35 (2.94) | 4.08 (1.95)

2. Primary Outcome: Time to Reach Maximum Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
hours
  Hydrocodone | 1.55 (0.71) | 3.38 (1.58) | 1.39 (1.22) | 3.09 (1.89)
  Acetaminophen | 0.91 (0.44) | 2.84 (1.49) | 0.80 (0.55) | 2.64 (1.44)
  Promethazine (Number of Participants=19,19,20,19) | 4.35 (1.37) | 5.24 (2.37) | 4.90 (1.72) | 6.45 (4.59)

3. Primary Outcome: Last Quantifiable Drug Concentration (Clast) Determined Directly From Individual Concentration-time Data
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
ng/mL
  Hydrocodone | 0.556 (0.354) | 0.523 (0.412) | 0.465 (0.315) | 0.527 (0.424)
  Acetaminophen | 0.0741 (0.0297) | 0.0917 (0.0378) | 0.0724 (0.0291) | 0.0907 (0.0428)
  Promethazine (Number of Participants=19,19,20,19) | 0.611 (0.936) | 0.586 (1.04) | 0.574 (0.829) | 0.701 (0.912)

4. Primary Outcome: Time of the Last Quantifiable Concentration (Tlast)
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
Hours
  Hydrocodone | 27.80 (8.99) | 31.21 (11.28) | 28.81 (9.84) | 31.58 (11.46)
  Acetaminophen | 23.38 (2.76) | 24.01 (0.04) | 23.41 (2.69) | 24.01 (0.02)
  Promethazine (Number of Participants=19,19,20,19) | 46.76 (5.51) | 46.77 (5.52) | 46.81 (5.37) | 46.74 (5.51)

5. Primary Outcome: Observed Elimination Rate Constant (λz)
Description: Estimated by linear regression through at least three data points in the terminal phase of the log concentration-time profile
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h-1
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h-1
  Hydrocodone | 0.1468 (0.0293) | 0.1373 (0.0258) | 0.1415 (0.0292) | 0.1371 (0.0271)
  Acetaminophen | 0.1577 (0.0310) | 0.1359 (0.0223) | 0.1600 (0.0355) | 0.1412 (0.0218)
  Promethazine (Number of Participants=19,18,20,18) | 0.0429 (0.0129) | 0.0451 (0.0451) | 0.0422 (0.0120) | 0.0458 (0.0145)

6. Primary Outcome: Observed Terminal Elimination Half-life (T1/2)
Description: Calculated as: T1/2 = ln(2)/λz
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
hours
  Hydrocodone | 4.93 (1.11) | 5.22 (0.99) | 5.13 (1.18) | 5.26 (1.08)
  Acetaminophen | 4.59 (1.06) | 5.22 (0.79) | 4.52 (0.93) | 5.03 (0.86)
  Promethazine (Number of Participants=19,18,20,18) | 17.49 (5.21) | 15.95 (3.04) | 17.77 (5.57) | 16.24 (4.09)

7. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC0-0.25) for Hydrocodone and Promethazine
Description: AUC0-0.25 measured by Linear Trapezoidal with Linear Interpolation method.
Time Frame: 0 (pre-dose) to 0.25 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 0.08870 (0.1318) | 0.03786 (0.1269) | 0.1219 (0.2151) | 0.02250 (0.04577)
  Promethazine (Number of Participants=19,19,20,19) | 0.01086 (0.03169) | 0.003941 (0.01413) | 0.006288 (0.02608) | 0.002612 (0.01138)

8. Primary Outcome: AUC0-0.50 for Hydrocodone and Promethazine
Description: AUC0-0.50 measured by Linear Trapezoidal with Linear Interpolation method.
Time Frame: 0 (pre-dose) to 0.5 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 0.9532 (0.9498) | 0.2566 (0.6382) | 1.280 (1.271) | 0.3163 (0.4305)
  Promethazine (Number of Participants=19,19,20,19) | 0.03535 (0.06239) | 0.01570 (0.03508) | 0.02692 (0.06096) | 0.01220 (0.02452)

9. Primary Outcome: AUC0-0.75 for Hydrocodone and Promethazine
Description: AUC0-0.75 measured by Linear Trapezoidal with Linear Interpolation method.
Time Frame: 0 (Pre-dose) to 0.75 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 3.194 (2.379) | 0.8759 (1.645) | 4.027 (3.092) | 1.276 (1.629)
  Promethazine (Number of Participants=19,19,20,19) | 0.1108 (0.1090) | 0.05549 (0.08128) | 0.09690 (0.1478) | 0.04610 (0.06227)

10. Primary Outcome: AUC0-1.0 for Hydrocodone and Promethazine
Description: AUC0-1.0 measured by Linear Trapezoidal with Linear Interpolation method.
Time Frame: 0 (pre-dose) to 1.0 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 6.383 (3.637) | 2.046 (3.244) | 7.524 (4.678) | 2.722 (3.329)
  Promethazine (Number of Participants=19,19,20,19) | 0.2578 (0.1999) | 0.1457 (0.1649) | 0.2311 (0.3055) | 0.1109 (0.1471)

11. Primary Outcome: AUC0-1.5 for Hydrocodone and Promethazine
Description: AUC0-1.5 measured by Linear Trapezoidal with Linear Interpolation method.
Time Frame: 0 (pre-dose) to 1.5 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 14.33 (4.971) | 5.782 (7.049) | 14.95 (6.822) | 6.424 (6.742)
  Promethazine (Number of Participants=19,19,20,19) | 0.8524 (0.5410) | 0.5573 (0.4798) | 0.7330 (0.8395) | 0.3239 (0.3643)

12. Primary Outcome: AUC0-2.0 for Hydrocodone and Promethazine
Description: AUC0-2.0 measured by Linear Trapezoidal with Linear Interpolation method.
Time Frame: 0 (pre-dose) to 2 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 23.21 (6.240) | 10.95 (10.34) | 22.53 (8.183) | 11.04 (10.12)
  Promethazine (Number of Participants=19,19,20,19) | 1.938 (1.318) | 1.267 (0.9936) | 1.583 (1.689) | 0.6735 (0.6328)

13. Primary Outcome: AUC0-4.0 for Hydrocodone and Promethazine
Description: AUC0-4.0 measured by Linear Trapezoidal with Linear Interpolation method.
Time Frame: 0 (pre-dose) to 4 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 54.04 (13.77) | 38.97 (18.47) | 48.35 (12.87) | 35.14 (17.97)
  Promethazine (Number of Participants=19,19,20,19) | 9.124 (6.271) | 5.943 (3.676) | 7.101 (6.159) | 4.045 (2.497)

14. Primary Outcome: Area Under the Plasma Concentration-time (AUClast) Curve From Time-zero to the Time of the Last Quantifiable Concentration
Description: Calculated using the linear trapezoidal rule
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 146.2 (56.77) | 151.9 (58.79) | 130.9 (47.94) | 148.5 (56.84)
  Acetaminophen | 19.19 (5.661) | 17.85 (4.621) | 18.69 (5.186) | 17.85 (4.742)
  Promethazine (Number of Participants=19,19,20,19) | 75.69 (78.87) | 66.63 (67.37) | 68.54 (63.24) | 74.76 (57.53)

15. Primary Outcome: Area Under the Concentration-time (AUCinf) Curve From Time-zero Extrapolated to Infinity
Description: Calculated as:
  AUCinf = AUClast + Clast/λz
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
h*ng/mL
  Hydrocodone | 150.2 (57.30) | 155.8 (58.75) | 134.3 (48.20) | 152.4 (56.83)
  Promethazine (Number of Participants=19,18,20,18) | 96.92 (119.5) | 60.72 (29.74) | 88.53 (100.3) | 84.13 (76.72)

16. Primary Outcome: Percentage of AUCinf [AUCExtrap (%)] Based on Extrapolation
Description: Calculated as:
  AUCExtrap (%) = (AUC0-inf - AUC0-last)/AUC0-inf *100
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours post-dose
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage of AUCExtrap
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Number analyzed (Participants) | 19 | 20 | 20 | 19
Percentage of AUCExtrap
  Hydrocodone | 2.72 (1.72) | 2.68 (1.97) | 2.65 (1.78) | 2.71 (2.06)
  Promethazine (Number of Participants=19,18,20,18) | 14.35 (7.03) | 13.54 (4.64) | 15.15 (7.86) | 14.56 (6.28)

ADVERSE EVENTS:
Time Frame: Up to day 72
Arm/Group | Treatment A: CL-108 (Fasted) | Treatment B: CL-108 (Fed) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 3/19 | 11/20 | 20/20 | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: CL-108 (Fasted) (N=19) | Treatment B: CL-108 (Fed) (N=20) | Treatment C: Vicoprofen, Ultracet and Phenergan (Fasted) (N=20) | Treatment D: Vicoprofen, Ultracet and Phenergan (Fed) (N=19)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 4 | 0
Oral pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 2 | 2
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 2 | 3 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No